CLINICAL TRIAL: NCT03240822
Title: Vascularized Composite Allotransplantation (VCA) for Devastating Penile and Concomitant Genital Trauma
Brief Title: Human Penile Tissue Allotransplantation for Devastating Penile and Concomitant Genital Trauma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027539
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-07

CONDITIONS: Urologic Injuries; Genital Diseases, Male; Amputation
Keywords: Penile Trauma; Allotransplantation; Vascularized Composite Allotransplantation; VCA; Genital Trauma; Penile Transplantation; Amputation; Penile Injury
MeSH Terms: conditions — Genital Diseases, Male | interventions — Antibodies, Monoclonal; Tacrolimus

STUDY DESIGN:
Intervention Model Description: All subjects receive transplant and immunosuppression therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Penile Allotransplant and Immunosuppression Treatment (Experimental): Penile transplantation with monoclonal antibody induction therapy of humanized anti CD52 followed by donor bone marrow infusion and tacrolimus monotherapy.
  Interventions: Procedure: Penile Transplant; Biological: Monoclonal Antibody (Humanized Anti-CD52); Drug: Tacrolimus

INTERVENTIONS:
Procedure: Penile Transplant — Penile Allotransplantation
Biological: Monoclonal Antibody (Humanized Anti-CD52)
Drug: Tacrolimus

SUMMARY:
This is a 4-year, non-randomized, single center, patient self-controlled, clinical trial (though enrolled subjects will be followed for life as are all transplant patients) for patients seeking allotransplantation of the male external genitalia (MEG), or penile tissue, as a feasible reconstructive strategy for the treatment of devastating and irreversible injuries to the genitalia. In addition to receiving penile allotransplantation and post-operative monitoring and support, enrolled patients will receive an innovative and clinically proven immunomodulatory protocol that combines lymphocyte depletion of the recipient with donor bone marrow cell infusion. Patients will be treated with lymphocyte depleting induction therapy, donor bone marrow cell infusion and tacrolimus. After the first year, maintenance immunosuppression will be modified gradually and cautiously (tapered dose reduction or spaced frequency dosing of tacrolimus) in selected patients based on a critical evaluation of clinical and immunologic outcomes. Outcomes will include but not be limited to functional metrics (sensation, erection, voiding), psychosocial (body integrity, adaptation to transplant) and health related quality of life (HRQOL) measures.

DETAILED DESCRIPTION:
Initial treatment with an antibody targeting recipient immune cells followed by triple-drug maintenance therapy represents the current standard in clinical VCA. Our protocol is different from the existing conventional drug treatments used in MEG allotransplantation in that it combines donor bone marrow infusion with an immunosuppression sparing protocol. The primary goal of this pilot clinical trial is to determine the feasibility of using allogeneic penile tissue to repair/replace irreversibly damaged external genitalia. Enrolled and transplanted subjects will be followed for their lifetime as a transplant patient.

ELIGIBILITY:
Inclusion Criteria: For Recipients

1. Male
2. 18-40 years
3. Irreversible and devastating genitalia damage not amenable to conventional reconstruction.
4. Patent main vessels leading into the remaining penile stump, as confirmed by angiography.
5. Adequate penile stump (> 2.5cm) to facilitate placement of a tourniquet, debridement of the distal portion and sufficient distal mobilization of the structures requiring anastomosis
6. Eligible for long term standard of care coverage

Exclusion Criteria: For Recipients

1. Documented history of:

   1. cancer
   2. renal impairment
   3. hepatic disorders
   4. neurologic disorders (sensory or motor function deficits)
   5. severe scarring with poor host tissue bed
   6. penile resection or implant surgery
   7. diabetes
   8. hypertension
   9. hyperlipidemia
   10. coronary artery disease
   11. untreated genital cancer
   12. HIV, Hepatitis B or C, or any infectious disease
   13. erectile dysfunction
   14. Peyronie's disease
   15. urethral stricture disease
   16. balanitis
   17. xerotica obliterans
   18. pelvic embolization
   19. pelvic radiation
   20. untreated hypogonadism
   21. prior prostate surgery
   22. recurrent urinary tract infections (UTIs)
   23. nephrolithiasis
   24. connective tissue disease or collagen disease
   25. lipopolysaccharidosis or amyloidosis
2. Use of 5-alpha-reductase inhibitors
3. External signs, sequelae or positive serology of sexually transmitted disease (including HPV)
4. Active UTI, stones, urethral edema and other pathology that prevents urethral anastomosis
5. Current or past substance abuse
6. Current or past smoker (within past 3 months)
7. Use of any medications known to cause vasoconstriction
8. Psychiatric illness or psychological problems, or deemed unsuitable on psychiatric evaluation
9. Any condition that may prevent transplantation (positive cross match, high panel reactive antibody (PRA), etc.)
10. Uncontrolled bleeding disorder, platelet count > 50,000, hemophilia or any other inherited coagulopathy or need to routinely receive blood products for bleeding disorders
11. Concurrent participation in any other clinical investigation during the period of this investigation
12. Inability to undergo leukapheresis
13. Inability to participate in all necessary study activities due to physical or mental limitations
14. Inability or unwillingness to return for all required follow-up visits.
15. Inability or unwillingness to sign the patient informed consent document.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a male, penile transplantation study.
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Need for Immunosuppressive drug therapy | 6 months
  The amount of immunosuppressive drug therapy will be recorded.

SECONDARY OUTCOMES:
erectile function | 6 months
  This will be assessed following intracorporal injection of vaso-active agents, such as prostaglandin, phentolamine, papaverine, or some mixture of these drugs (i.e. Trimix). and through high-resolution duplex Doppler ultrasonography
Assessment of sensory return and sensory thresholds | 6 months
  This will be accomplished by penile biothesiometry
Determination of hemodynamic status | 6 months
  Dynamic infusion pharmaco-cavernosometry and cavernosography will be utilized to better understand these changes
The Reintegration to Normal Living (RNL) Index | 6 months
  The RNL is an 11-item questionnaire that asks how a person manages activities, roles, and relationships on a day-to-day basis.
The Situational Inventory of Body-Image Dysphoria (SIBID) | 6 months
  The SIBID is a multidimensional body-image survey assessment of people's negative body-image emotions in everyday situations and physical experiences.
The Function and Body Image Survey | 6 months
  This survey consists of six open-ended questions regarding personal thoughts, opinions, and experiences about the transplant, and the individual's current functional abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Atala, MD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No